CLINICAL TRIAL: NCT05441384
Title: It Is Time to Address Fear of Cancer Recurrence in the Family Caregiver: Adaptation, Feasibility, and Acceptability Study of an Online Version of the Fear Of Recurrence Therapy
Brief Title: It's Time to Address Fear of Cancer Recurrence in Family Caregivers: Online Version of the Fear Of Recurrence Therapy
Acronym: FC-FORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Sophie Lebel, Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-05-20-5584
Record Dates: First submitted 2022-06-15; First posted 2022-07-01 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Cancer; Caregiver; CBT; Fear Cancer
Keywords: Pilot Study; Group Therapy; Virtual
MeSH Terms: conditions — Neoplasms; Pathophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT/Existential Group Therapy for Fear of Cancer Recurrence (Experimental): Participants will receive 7 weekly group therapy sessions consisting of psychoeducation on fear of cancer recurrence, relaxation training, CBT, and evidenced-based tips to decrease avoidance and anxiety surrounding fear of cancer recurrence.
  Interventions: Behavioral: Family Caregiver - Fear Of Recurrence Therapy (FC-FORT)
- Wait-list Control Group (No Intervention): Participants assigned to this arm wait about 3-months to receive the intervention.

INTERVENTIONS:
Behavioral: Family Caregiver - Fear Of Recurrence Therapy (FC-FORT) — 7 weekly sessions of 90-120 minutes each. During the 7 weeks, participants will be asked to participate in activities, participate in group discussions, and complete homework assignments.
  Arms: CBT/Existential Group Therapy for Fear of Cancer Recurrence

SUMMARY:
Fear of cancer recurrence (FCR) is common, persistent, and is associated with negative outcomes. Studies show that family caregivers (FC) of cancer patients experience equal or greater levels of FCR than patients themselves. In the past 5 years, several interventions have demonstrated their ability to reduce FCR among cancer patients, including a group intervention called Fear of Recurrence Therapy (FORT). However, none have ever been adapted and offered to caregivers. The goals of the proposed study are to demonstrate 1) that a newly adapted intervention of FORT (FC-FORT) is feasible (i.e., participant recruitment, attendance and participation) and acceptable (i.e., FC satisfaction of the intervention) for a larger study, and 2) the clinical implications of FC- FORT on FCR and quality of life. An advisory board composed of researchers, therapists, and FC was created to adapt FORT for FC and to an online format. FC and therapists are currently being recruited to conduct a usability study of the newly adapted FC-FORT. They will be asked to complete a session feedback questionnaire after each session and to take part in an exit interview. The content of these will be summarized back to the advisory board in order to further refine FC-FORT. Following a successful usability study, FC-FORT will be given to four groups of nine new FC (pilot study). Participants will be recruited directly by clinicians and by outreach mailout efforts. They will complete a questionnaire package before and after the intervention, as well as at a three month follow up. The proposed study is needed to determine if an already developed FCR intervention can be adapted to family caregivers and if it can be successfully pilot tested. This will help bridge an important gap in bringing evidence-based care to caregivers who have never been offered help before for their FCR. The proposed project will also allow to further feasibility and acceptability of E-Health interventions.

DETAILED DESCRIPTION:
Usability Study

6-8 female family caregivers will be recruited to conduct a usability study of this first version of FC-FORT. Participants will be recruited through the University of Ottawa, the Princess Margaret Cancer Centre, community partners and social media. Two therapists with extensive experience with online support groups to conduct the sessions will be recruited to conduct the groups. Therapist competency to administer FC-FORT will be determined by registered professionals in counselling or psychotherapy, at least 5 years of experience in psychosocial oncology, and having led at least one group. These therapists will receive an online training from the principal investigators before starting the usability study. Interested family caregivers will contact the research coordinator, via telephone or email, to be screened for eligibility and to complete the consent forms. All eligible participants will attend a one-on-one pre-therapy meeting to prepare them for the group work (i.e.: review expectations and assess whether group work is appropriate for the participant) and complete the 7-week FC-FORT intervention. Before starting the intervention, participants will receive a standardized manual describing each session's activities and assignments. After each of the seven sessions, the therapists and the participants will be asked to complete a short session feedback questionnaire, via Qualtrics, to assess the usefulness, usability, desirability, value, accessibility, and credibility of the session, as well as about participants' impressions of the online format and features, and the general readiness of the session for end users. Brief videoconference or telephone exit interviews will be conducted post-intervention with both the participating family caregivers and the therapists. The content of these interviews and questionnaires will be summarized and present it back to the project's advisory board in order to further refine the FC-FORT content and format.

Pilot Study

36 family caregivers will be recruited to participate in the study. Additionally, 3 therapists with extensive online support group experience to conduct the FC-FORT videoconference therapy sessions. Therapist competency to administer FC-FORT will be determined by registered professionals in counselling or psychotherapy, at least 5 years of experience in psychosocial oncology, and having led at least one group. Interested family caregivers will contact the research coordinator, via telephone or email, to be screened for eligibility and to complete the consent forms. This pilot study will serve as a first step in potential sample size calculations and recruitment times. For this pilot study, active recruitment will last for a period of 15 months during which 36 FC are aimed to be recruited in order to create 4 groups of 9 participants (2 intervention conditions and 2 WLCG). Feasibility of recruitement for the larger RCT will be determined using these critera: 1) If during our recruitment period less than 18 participants, recruitement for a larger RCT, using our current recruitment strategies, will be deemed not feasible, 2) If between 18 and 25 participants are recruited, then a larger multicentre approach for recruitment will be considered, 3) If recruit 25 participants or more, recruitement for a larger RCT, using our current methods, will be deemed feasible. The sample size will be reevaluated for the larger RCT based on the results from this pilot study.

FC-FORT consists of 7 consecutive weekly group sessions of 90-120 minutes each offered through videoconference and weekly assigned homework. FC-FORT is therapist led, however participants will receive a workbook where they can follow along, take notes, and complete the exercises and the homework assignments. The overall aim of FC-FORT is to guide FC towards a more manageable level of worry and fear of recurrence. The key goals are to: 1) distinguish worrisome symptoms from benign ones; 2) identify FCR triggers and inappropriate coping strategies; 3) facilitate the learning and use of new coping strategies, such as relaxation techniques, cognitive restructuring, communication strategies and the use of self-care; 4) increase tolerance for uncertainty; 5) promote emotional expression of specific fears that underlie FCR; and 6) re-examine life priorities and set realistic goals for the future. Each session is composed of exercices where participants have to answer questions, share with the group or watch videos. Furthermore, homework is assigned after each session to be completed before next week's session. Eligible participants will attend a one-on-one pre-therapy meeting with a study therapist to prepare them for the group work (i.e.: review expectations and assess whether group work is appropriate for the participant) and complete the 7-week FC-FORT intervention. Membership will be closed once groups are formed and the sessions have started to enhance group cohesiveness and consistency. Before starting the intervention, participants will receive a standardized manual describing each session's activities and assignments. All participants (including those in the wait list control group) will complete a questionnaire package pre intervention, post intervention, and at a three month follow up via Qualtrics. Additionally, participants will be asked to complete post session measures, namely the Working Alliance Inventory - Revised Short Form as well as the Group Cohesiveness Scale after the 1st, 4th and 7th sessions.

Therapist Training and Supervision.

To enhance therapist adherence to treatment, the therapists recruited for the study will be provided with a standardized FC-FORT manual and will be trained by the research psychologists through an online training. The research team will review the video of each session and the principal investigator will provide weekly 30-minute supervision to the therapists. Furthermore, the study will use an updated version of the fidelity checklist that was used to evaluate adherence during the previous FORT studies. If adherence is less than 80% on any session, the research team will provide additional over-the-telephone feedback to the therapists running the group. This approach to monitoring treatment integrity and fidelity has been successful in previous FORT studies.

Qualitative Assessment.

To gain further insights about the feasibility, acceptability, and potential clinical significance of the FC-FORT, all study participants will be asked to complete semi structured interviews. This will enable a holistic understanding of their experience of FC-FORT, elucidate key intervention processes, and identify additional secondary outcomes. Lastly, the research coordinator will attempt to interview participants who dropped out of the intervention, to understand any hindering factors. Consenting participants will be asked to complete a semi structured interview (30-60 minutes) about their experience of the intervention through videoconferencing.

Randomization

This study will use a mixed method randomized control trial design using a waitlist control group and 3 months follow up, with 18 participants per condition. To minimize attrition associated with waiting to enroll participants, block randomization will be used. Specifically, a list of 4 blocks with equal numbers of intervention (I) and wait list control (WLCG) groups (e.g. I-I-WLCG-WLCG; I-WLCG-WLCG-I, etc.) will be randomly created. Once the first 9 participants have been recruited, they will be assigned to whichever group came up first on the list. The next 9 participants will be assigned to the next group on the generated list until all 4 groups have been completed. Participants assigned to the WLCG will be offered the intervention after the 3-month period. To limit bias, each of the 4 blocks of the list will be in separate sealed envelopes that will be opened one at a time after 9 participants have been recruited.

Minimizing Dropouts and Attrition

To maximize attendance, as in our prior research, participants will be told during informed consent procedures about the importance of attending all 7 sessions to ensure benefit from the intervention. Participants will receive two email reminders about each upcoming session, along with "homework" and session pre-reading materials. They will be asked to inform group therapists if they are to be absent. For participants who miss a session, they will be offered one individual videoconference make-up session for their first missed session before the next group; they will not be offered subsequent make-up sessions for additional missed sessions to decrease the risk that this would encourage those who prefer individualized attention to miss group sessions. Participants who miss more than two sessions will be asked to stop the intervention and restart with the next available group. This approach was successfully tested in previous FORT studies. To minimize differential attrition from the WLCG participants, participants will be emailed monthly with an update about the wait time.

Feasibility and Acceptability Criteria.

The following criteria will be used to assess the feasibility and acceptability of FC-FORT: 1) ability to recruit 36 FC in 15 months; 2) ability to randomize these 36 FC; 3) ability to deliver FC-FORT to 27 FC in 15 months (25% dropout rate); 4) 80% completion of 6 out of the 7 sessions; 5) complete measures for 90% of participants; 6) ability to deliver FC-FORT as intended as measured by a fidelity rating of above 80% on 75% of reviewed sessions; and 7) FC satisfactory ratings >than 80% in terms of its content, therapists, and mode of delivery.

Quantitative analysis.

Descriptive statistics will be used to report on FCR outcomes. A linear mixed-effect model analyses will be done on the secondary outcome measures pre- and post-intervention and at the 3-month follow-up. All analyses will use both an intent-to-treat and per protocol approaches. Known extraneous variables that could influence FCR (e.g., age, education, income, cancer stage) will be measured and control for, and monitor for participants' use of any additional psychological support at each data-collection time-points. Dependence of the group data will be analyzed with an intraclass correlation coefficient (p) using a multilevel model.

Qualitative Analysis.

Conventional content analysis will be used to analyse the qualitative data. Interviews will be audiotaped, transcribed verbatim, and managed using the qualitative software program NVivo. Transcripts will be systematically coded into anticipated (e.g., motivations to participate, benefits of participation) and emergent codes. This is an iterative process whereby an initial set of themes are coded, applied to new transcripts, and revised to adjust for new information, until no new codes emerge. Double coding of 80% of the interviews will be done by the research assistant. These codes will then be sorted into subcategories (ideally between 10 to 15).

ELIGIBILITY:
Inclusion Criteria:

* Female adult FC caring for an adult cancer survivor of any type of cancer type, stages I-III, who has completed treatments and has not had a recurrence of their cancer;
* A score of 13 or greater on the Fear of Cancer Recurrence Inventory-Short Form (range 0-36), suggesting clinical levels of FCR;
* Access to a computer and stable internet connection;
* Living in Canada.

Exclusion Criteria:

* Individuals who do not identify as female;
* Family caregiver of a pediatric cancer survivor;
* Non-English speaking;
* Currently participating in another therapist-led psychosocial support group or a peer-led support group;
* Individuals with unmanaged/undermanaged mental health disorder judged to be clinically contra-indicated and/or likely to affect the group work.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals identifying as female.
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in baseline fear of cancer recurrence after intervention | Changes in baseline fear of cancer recurrence 7 weeks after the start of the intervention
  Fear of Cancer Recurrence Inventory - Short Form (FCR-SF), range from 0-36 with higher scores indicating high levels of fear of cancer recurrence
Changes in baseline fear of cancer recurrence at three months | Changes in baseline fear of cancer recurrence 3 months after the start of the intervention
  Fear of Cancer Recurrence Inventory - Short Form (FCR-SF), range from 0-36 with higher scores indicating high levels of fear of cancer recurrence

SECONDARY OUTCOMES:
Changes in Baseline Intolerance of Uncertainty Scale at 7 Weeks | Changes in baseline Intolerance of Uncertainty Scale after 7 weeks of the intervention
  Intolerance of Uncertainty Scale - Short Form (IUS-SF), range from 12-60 with higher scores indicating high levels of intolerance of uncertainty
Changes in Baseline Intolerance of Uncertainty Scale at 3 Months | Changes in baseline Intolerance of Uncertainty Scale at 3 month after the completion of the intervention
  Intolerance of Uncertainty Scale - Short Form (IUS-SF), range from 12-60 with higher scores indicating high levels of intolerance of uncertainty
Changes in baseline Uncertainty in Illness at 7 weeks | Changes in baseline Intolerance of Uncertainty Scale after 7 weeks of the intervention
  Mishel Uncertainty in Illness Scale Short-Form, range from 5-25 with higher scores indicating high levels of uncertainty in illness
Changes in baseline Uncertainty in Illness at 3 months | Changes in baseline Intolerance of Uncertainty Scale at 3 month after the completion of the intervention
  Mishel Uncertainty in Illness Scale Short-Form, range from 5-25 with higher scores indicating high levels of uncertainty in illness
Changes in baseline Positive Beliefs About Worrying at 7 weeks | Changes in baseline Positive Beliefs About Worrying after 7 weeks of the intervention
  Why Worry Questionnaire (WWQ), range from 13-65 with higher scores indicating more positive beliefs about worrying
Changes in baseline Positive Beliefs About Worrying at 3 months | Changes in baseline Positive Beliefs About Worrying at 3 month after the completion of the intervention
  Why Worry Questionnaire (WWQ), range from 13-65 with higher scores indicating more positive beliefs about worrying
Changes in baseline avoidance at 7 weeks | Changes in baseline avoidance after 7 weeks of the intervention
  Cognitive Avoidance Questionnaire (CAQ), range from 25-125 with higher scores indicating higher use of avoidance as a coping strategy
Changes in baseline avoidance at 3 months | Changes in baseline Avoidance at 3 month after the completion of the intervention
  Cognitive Avoidance Questionnaire (CAQ), range from 25-125 with higher scores indicating higher use of avoidance as a coping strategy
Changes in baseline Protective Buffering at 7 weeks | Changes in baseline protective buffering after 7 weeks of the intervention
  Protective Buffering Scale (PBS), range from 10-50 with higher scores indicating high levels of protective buffering
Changes in baseline Protective Buffering at 3 months | Changes in baseline protective buffering at 3 month after the completion of the intervention
  Protective Buffering Scale (PBS), range from 10-50 with higher scores indicating high levels of protective buffering
Changes in Therapeutic Alliance at weeks 1, 4, and 7 | Changes in baseline therapeutic alliance through study completing (at weeks 1, 4 and 7)
  Working Alliance Inventory - Revised Short Form (WAI-R-SF), Range from 12-60 with higher scores indicating a stronger therapeutic alliance
Changes in Group Cohesion at weeks 1, 4, and 7 | Changes in baseline group cohesion through study completing (at weeks 1, 4 and 7)
  Group Cohesiveness Scale (GCS), Range from 7-35 with higher score indicating a stronger group cohesion

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lebel, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maheu C, Lebel S, Courbasson C, Lefebvre M, Singh M, Bernstein LJ, Muraca L, Benea A, Jolicoeur L, Harris C, Ramanakumar AV, Ferguson S, Sidani S. Protocol of a randomized controlled trial of the fear of recurrence therapy (FORT) intervention for women with breast or gynecological cancer. BMC Cancer. 2016 Apr 25;16:291. doi: 10.1186/s12885-016-2326-x. PMID 27112319
- [Background] Moran C, Tomei C, Lefebvre M, Harris C, Maheu C, Lebel S. An exploratory study of the worst-case scenario exercise as an exposure treatment for fear of cancer recurrence. Support Care Cancer. 2017 May;25(5):1373-1375. doi: 10.1007/s00520-017-3600-4. Epub 2017 Feb 2. PMID 28150044
- [Background] Maheu C, Lebel S, Tomei C, Singh M, Esplen MJ. Breast and ovarian cancer survivors' experience of participating in a cognitive-existential group intervention addressing fear of cancer recurrence. Eur J Oncol Nurs. 2015 Aug;19(4):433-40. doi: 10.1016/j.ejon.2014.12.003. Epub 2014 Dec 30. PMID 25555320
- [Background] Tomei C, Lebel S, Maheu C, Lefebvre M, Harris C. Examining the preliminary efficacy of an intervention for fear of cancer recurrence in female cancer survivors: a randomized controlled clinical trial pilot study. Support Care Cancer. 2018 Aug;26(8):2751-2762. doi: 10.1007/s00520-018-4097-1. Epub 2018 Mar 2. PMID 29500582
- [Derived] Lamarche J, Nissim R, Avery J, Wong J, Maheu C, Lambert SD, Laizner AM, Jones J, Esplen MJ, Lebel S. It is Time to Address Fear of Cancer Recurrence in Family Caregivers: Feasibility and Acceptability of a Randomized Pilot Study of the Family Caregiver Version of the Fear of Recurrence Therapy (FC-FORT). Psychooncology. 2025 Feb;34(2):e70084. doi: 10.1002/pon.70084. PMID 39887474
- [Derived] Lamarche J, Nissim R, Avery J, Wong J, Maheu C, Lambert SD, Laizner AM, Jones J, Esplen MJ, Lebel S. It is time to address fear of cancer recurrence in family caregivers: protocol for the feasibility and acceptability of a randomized pilot study of the online version of the Family Caregiver-Fear Of Recurrence Therapy (FC-FORT). Pilot Feasibility Stud. 2024 Nov 19;10(1):143. doi: 10.1186/s40814-024-01567-4. PMID 39563465
- See also: Related Info — https://socialsciences.uottawa.ca/psychosocial-oncology-laboratory/fort-0